CLINICAL TRIAL: NCT04283487
Title: Brain and Gut Responses to Intragastric Administration of FODMAPs in Healthy Subjects and Patients With Irritable Bowel Syndrome
Acronym: FODMAPs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: FODMAP2
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAP; Irritable bowel syndrome; brain-gut axis; fMRI; abdominal MR
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Fructans; Glucose; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, crossover
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fructans solution (Experimental): Fructans (FODMAP) are oligosaccharides containing fructose chains. Since the human body lacks hydrolases to break down these saccharides, fructans are poorly absorbed molecules in everybody.The fructans solution used in this study is 500 ml water containing 40g fructans
  Interventions: Dietary Supplement: Fructans
- Glucose solution (Active Comparator): Glucose is a carbohydrate that is not classified as FODMAP, and is therefore used as a positive control in this study. The glucose solution used in this study is 500 ml water containing 40g glucose.
  Interventions: Dietary Supplement: Glucose
- Saline solution (Placebo Comparator): The saline solution does't contain any sugar and used in this study is 500ml 0.9% normal saline.
  Interventions: Dietary Supplement: Saline

INTERVENTIONS:
Dietary Supplement: Fructans — 500ml 0.9% normal saline containing 40g fructans
  Arms: Fructans solution
Dietary Supplement: Glucose — 500ml 0.9% normal saline containing 40g glucose
  Arms: Glucose solution
Dietary Supplement: Saline — 500ml 0.9% normal saline
  Arms: Saline solution

SUMMARY:
Low fermentable oligo-, di- and monosaccharides and polyols (FODMAPs) diet is taken as a possible strategy to improve symptoms in IBS patients. However, the gut-brain signalling mechanisms underlying this observation remain poorly understood. In this study, the investigators aim to study the brain mechanisms underlying the effect of intragastric administration of one specific FODMAP (fructans) on gastrointestinal and non- gastrointestinal symptom responses, changes in gut physiology(morphology of the gut, water content and intestinal motility), and to relate the findings to changes in gastrointestinal peptides. Intragastric administration of three different solutions will be given after an overnight fast: one FODMAP solution (fructans), a positive control (glucose) and a negative control (saline). The whole procedure consists of a functional magnetic resonance imaging (fMRI) and abdominal MRI examination, and will take approximately four hours. The participants will undergo the fMRI for one hour for assessing brain activity, during which blood samples will be collected. The abdominal MRI will be performed at 1-hour interval for three hours to assess pre and post stimulated changes in gut physiology, specifically the morphology of the gut water content and pan-intestinal motility. During the whole procedure, questionnaires for assessing the gastrointestinal symptoms and emotional state will be collected. The investigators hypothesise that fructans induce distension and increased sensations of pain, cramps and flatulence in the IBS group more than the HC. Furthermore, this will be associated with increased activation of pain-responsive brain regions in IBS compared to HC, which will be mediated by differential changes in gut peptide levels (↓ in orexigenic and ↑ in anorexigenic hormones).

DETAILED DESCRIPTION:
In this study, the investigators aim to study the brain mechanisms underlying the effect of intragastric administration of one specific FODMAP (fructans) on gastrointestinal and non- gastrointestinal symptom responses, changes in gut physiology(morphology of the gut, water content and intestinal motility), and to relate the findings to changes in gastrointestinal peptides.

This is a randomised, double-blinded, crossover study. Eligible participants will come three times to the clinic after an overnight fast, for intragastric infusion of fructans (40g in 500 ml water), glucose(40g in 500ml water) or saline(0.9% 500ml normal saline). The infusions will be given in counterbalanced order and with a washout period of at least one week. Participants and investigators will be blinded to the nature of the test solution, which will be made by a colleague unrelated to the study. The order of the test solutions will be determined by a computer-generated list. All participants will be asked to follow the low FODMAP diet for the 24 hours prior to each study day. Participants will be asked to record their food intake during the day to check their FODMAP intakes were reduced.

To begin, the participants will have a nasogastric feeding tube placed and an intravenous cannula inserted in the non-dominant arm to facilitate repeated blood sampling. Fifteen minutes later, they will enter the MR scanner for a 5 minute adaptation period. Participants will complete visual analogue scales (VAS) on appetite-related sensations and GI symptoms and blood samples will be collected for gut peptide analysis. Current emotional state will be rated before and after scanning using the PANAS, and during scanning using the POMS. The abdominal MRI scan will begin after the adaption period and will take 10 minutes. Hereafter, brain scanning will be performed, starting with a baseline brain scanning period of 10 minutes. After the baseline scanning, 500 mL of one of the three solutions will be infused as the functional brain imaging begins (and continues for 50 minutes). The VAS ratings will be collected every 10 minutes and blood samples will be collected every 20 minutes for measuring of ghrelin, CCK, GLP-1, motilin, and PYY, insulin and glucose throughout the scan. At 60 minutes post-infusion, a 10 minute abdominal scan will be acquired. After that, the subject leaves the scanner and the catheter will be removed. The subject will remain at the facility for a 2 hour follow-up during which the VAS ratings will be collected every 30 minutes and an abdominal MRI will be performed at 120 minutes post infusion. After the last abdominal MRI scan is performed, the infusion tube will be removed and the participant can go home.

ELIGIBILITY:
Healthy volunteers:

Inclusion Criteria:

* No symptoms or history of gastrointestinal disease or disorder, other significant diseases
* Female
* Age 18 - 55 years
* Body Mass Index (BMI) of 19 - 28 kg/m2
* Stable body weight for at least 3 months prior to the start of the study
* Right-handed or ambi-dexter

Exclusion Criteria:

* Medical
* Abdominal or thoracic surgery. Exception: appendectomy
* Gastrointestinal, endocrine or neurological diseases
* Cardiovascular, respiratory, renal or urinary diseases
* Hypertension
* Food or drug allergies
* Anemia Psychiatric disorders
* Eating disorders
* Depressive disorders
* Anxiety disorders
* Psychotic disorders Medication use
* No regular medication affecting CNS or GI system (oral contraception accepted) Other
* Conditions that can interfere with functional magnetic resonance imaging (fMRI), e.g. cochlear implants, metal fragments or metal implants in the body, pacemaker, neural stimulator, …
* No history of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 14 units for woman per week)
* People who show abnormal eating behavior or have followed a gluten-free or low-FODMAP diet previously
* Pregnant or breastfeeding women
* Claustrophobia

IBS patients:

Inclusion Criteria:

* Meet the Rome IV criteria for irritable bowel syndrome (IBS)
* Patient has IBS of any subtype
* Female
* Age 18 - 55 years
* Body Mass Index (BMI) of 19 - 28 kg/m2
* Stable body weight for at least 3 months prior to the start of the study
* Right-handed or ambi-dexter

Exclusion Criteria:

General exclusion criteria for all subjects:

Medical

* Abdominal or thoracic surgery. Exception: appendectomy
* Gastrointestinal, endocrine or neurological diseases
* Cardiovascular, respiratory, renal or urinary diseases
* Hypertension
* Food or drug allergies
* Anemia Psychiatric disorders
* Eating disorders
* Depressive disorders
* Anxiety disorders
* Psychotic disorders Medication use
* No regular medication affecting CNS or GI system (oral contraception accepted)

Other

* Conditions that can interfere with functional magnetic resonance imaging (fMRI), e.g. cochlear implants, metal fragments or metal implants in the body, pacemaker, neural stimulator, …
* No history of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 14 units of alcohol per week)
* People who show abnormal eating behavior, or have followed a gluten-free or low-FODMAP diet previously
* Pregnant or breastfeeding women
* Claustrophobia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Change in brain activation patterns measured by fMRI | -10 min to 50 min
  change in blood oxygenation level dependent (BOLD) signal by fMRI

SECONDARY OUTCOMES:
Change in gastrointestinal symptom scores measured by VAS | -30 min to 180 min
  bloating, nausea, cramps, flatulence and abdominal pain
Change in state emotion score measured by validated questionnaire | -30 min to 180 min
  emotion score measured by POMS
Change in state emotion score measured by validated questionnaire | -30 min to 180 min
  emotion score measured by PANAS
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of ghrelin
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of CCK
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of GLP-1
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of motilin
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of PYY
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of insulin
Change in plasma levels of gut peptides | -20 min to 60 min
  Plasma levels of glucose
Change in gut physiology measured by abdominal MRI | -20 min to 180 min
  Gastric emptying and accommodation, antral and small bowel motility, water and gas content measured by abdominal MRI

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PHD, Principal Investigator — UZ Leuven / KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the reported results will be made available 3 months after publication for a period of 5 years after the publication date upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Deidentified individual participant data that underlie the reported results will be made available 3 months after publication for a period of 5 years after the publication date upon request.

REFERENCES:
- [Derived] Wu J, Masuy I, Biesiekierski JR, Fitzke HE, Parikh C, Schofield L, Shaikh H, Bhagwanani A, Aziz Q, Taylor SA, Tack J, Van Oudenhove L. Gut-brain axis dysfunction underlies FODMAP-induced symptom generation in irritable bowel syndrome. Aliment Pharmacol Ther. 2022 Mar;55(6):670-682. doi: 10.1111/apt.16812. Epub 2022 Feb 15. PMID 35166384